CLINICAL TRIAL: NCT00850187
Title: Treatment of Full-thickness Articular Cartilage Defects in the Knee of Patients With Autologous Bone-marrow Mesenchymal Stem Cells and Scaffold
Brief Title: Autologous Transplantation of Mesenchymal Stem Cells (MSCs) and Scaffold in Full-thickness Articular Cartilage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan - Bone - 001
Record Dates: First submitted 2009-02-21; First posted 2009-02-24 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2010-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee cartilage diseases
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone marrow mesenchymal stem cells (Experimental)
  Interventions: Biological: Bone marrow derived mesenchymal stem cells

INTERVENTIONS:
Biological: Bone marrow derived mesenchymal stem cells — Bone Marrow Aspiration A total volume of 300 ml bone marrow will be aspirated from the iliac crest and are cultured for mesenchymal stem cells

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Bone Marrow Mesenchymal stem cells (MSCs) mixed with collagen I scaffold in patient with Knee cartilage defects and osteoarthritis

DETAILED DESCRIPTION:
Articular cartilage defects have a weak potential for self-repair because of the reduced mitotic capacity of chondrocytes in vivo. Because some patients with articular cartilage defects may progress to osteoarthritis, such defects need to be repaired even though their exact natural course remains obscure. Traditional methods for repair, such as micro fracture, perforations, abrasion arthroplasty, have not produced consistent satisfactory long term clinical results. Transplantation of autologous bone marrow MSCs expanded in culture would be a promising approach in the repair of articular cartilage defects in human osteoarthritic knees. This method is clinically straightforward to perform because autologous cells can be readily harvested and expanded in culture without losing their capacity to differentiate into chondrocytes. The purpose of this study was to evaluate the clinical results obtained with autologous MSCs expanded in culture for the treatment of full-thickness chondral defects in human knee.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 60, inclusive
* Normal axial alignment
* Stable knee-previous ligament reconstruction, if stable
* Intact articular cartilage in posterior meniscal weight-bearing zone
* Ability to understand and willingness tosign consent from
* O.C.D or OA calgran classification II,III

Exclusion Criteria:

* Pregnant or lactating
* Inflammatory arthritis
* Oral steriod, methotrexate
* Unable to follow post-operative exercise regimen or return for evaluations

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Knee cartilage defects | 12 months

SECONDARY OUTCOMES:
pain | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid gourabi, PhD, Study Chair — Chief; Mohamadreza Baghaban Eslaminejad, PhD, Study Director — Scientific Board; Leila Taghiyar, Msc, Principal Investigator — Researcher
Locations (2):
- Iran (2):
  - Royan Institute, Tehran, Tehran Province
  - Royan Institute, Tehran

REFERENCES:
- See also: Related Info — http://www.royaninstitute.org